CLINICAL TRIAL: NCT05639283
Title: Primary Obstructive Megaureter Management in Eastern Interregional Area : Current Status and Perspectives
Brief Title: Primary Obstructive Megaureter Management in Eastern Interregional Area
Acronym: POMME
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7978
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Congenital Obstructive Megaureter
Keywords: Congenital obstructive megaureter; Urinary malformation; Ureterovesical junction; Hydronephrosis; Renal dysplasia
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital obstructive megaureter is a urinary malformation affecting the ureterovesical junction and causing obstruction to the flow of urine. It is the second most common cause of hydronephrosis. This malformation affects four times more boys than girls and is bilateral in 25% of cases. It is also associated with contralateral renal dysplasia in 15% of cases. The obstruction is linked to aperistalsis and hypertrophy of the circular muscle bundles and increased collagen 1 level. This malformation is accessible to antenatal screening from the second trimester. It falls within the scope of CAKUT and requires regular monitoring. Indeed, this uropathy can cause repeated pyelonephritis, kidney scarring and affected kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient (from 1 to 17 years old)
* Patient treated between January 2010 and December 2017 in one of the participating centers for an obstructive congenital mega-ureter
* Subject (and/or his parental authority) not having expressed, after information, his opposition to the reuse of his data for the purposes of this research

Exclusion Criteria:

* Subject (and/or his parental authority) having expressed, after information, his opposition to the reuse of his data for the purposes of this research

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient (from 1 to 17 years old) treated between January 2010 and December 2017 for an obstructive congenital mega-ureter
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Determine over the past seven years, the operability factors of patients aged 0 to 5 years regardless of the surgical technique used | Files analysed retrospectively from January 01, 2010 to December 31, 2017 will be examined
  This study aims to make a retrospective inventory and perspective on the management of congenital obstructive mega ureter

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie pédiatrique - CHU de Strasbourg - France, Strasbourg, France